CLINICAL TRIAL: NCT05128786
Title: A Phase I Trial to Assess Safety, Tolerability and Anti-tumor Activity of Autologous T Cell Modified Chimeric Antigen Receptor (CAR) (CCT301-38) in Patients With Relapsed or Refractory AXL Positive Sarcomas
Brief Title: CCT301-38 CAR-T in Patients With Relapsed or Refractory AXL Positive Sarcomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Adjustment of study strategy
Sponsor: Shanghai PerHum Therapeutics Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCT301-38-SAR
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2023-04

CONDITIONS: SAR
Keywords: AXL, CAR-T, CCT301-38, sarcoma; CAR-T; CCT301-38; sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCT301-38 (Experimental): To determine the safety, tolerability, DLT and MTD of CCT301-38 cell therapy in patients with AXL-positive relapsed or refractory sarcomas.
  Interventions: Biological: CCT301-38

INTERVENTIONS:
Biological: CCT301-38 — Blood will be collected from subjects to isolate peripheral blood mononuclear cells for the production of CCT301-38. Subjects will receive the conditioning chemotherapy regimen of cyclophosphamide and fludarabine for lymphodepletion followed by a single or multiple dose of CCT301-38 via intravenous injection.

SUMMARY:
This clinical study is to investigate the safety and tolerability of CCT301-38 CAR modified autologous T cells (CCT301-38) in subjects with relapsed or refractory AXL positive sarcomas

DETAILED DESCRIPTION:
This study is an open label, single-center Phase I dose escalation trial to assess the safety, tolerability, DLT and MTD of CCT301-38 cell therapy in patients with AXL positive relapsed or refractory sarcomas.

Subjects that meet inclusion criteria with positive AXL biopsy (IHC 1+ or greater in ≥50% tumor cells) will receive CCT301-38 according to the 3+3 dose escalation design.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with willingness to be in the study and follow all study procedures, and capable of providing informed consent
2. Male or female aged 18-70 years;
3. Patients with unresectable, locally advanced or metastatic relapse/refractory sarcomas that have failed at least the front line standard treatment confirmed by histology or cytology;
4. At least one measurable lesion, i.e. the length of non-lymph node lesions examined according to CT cross-sectional scanning or magnetic resonance imaging (MRI), or the short diameter of the lymph node lesions is ≥15 mm according to RECIST 1.1, and the FDG PET signal from the measurable lesion is > 3 SUV;
5. Tumors with AXL positive (IHC 1+ or greater) in ≥50% of all tumor cells. A new biopsy is required if the sample is over one year.
6. ECOG Performance Status 0-1;
7. Expected survival greater than 12 weeks;
8. Adequate organ and hematopoietic system functions to meet the following requirements:

   * Hemoglobin (HGB) s 90 g/L, no blood transfusions within two weeks;
   * White blood cell (WBC) count≥2.5×109/L；
   * Absolute Neutrophil Count (ANC) ≥1.5×109/L;
   * Platelet (PLT) count ≥80×109/L;
   * Total bilirubin (TBIL) ≤3.0ng/dL or ≤5 ULN;
   * ALT and AST ≤5 ULN; for liver metastasis, ALT and AST ≤5 ULN
   * Creatinine (Cr) ≤1.5 x ULN; or creatinine removal rate (CrCl) ≥50 mL/min;
9. PT: INR < 1.7 or extended PT to normal value < 4s
10. Normal language, recognition and consciousness assessed by investigator during screening phase;
11. Capable of receiving treatment and follow-up, including treatment in the clinical center;

Exclusion Criteria:

1. Females with pregnancy or in lactation period;
2. Subjects with active hepatitis B, or active hepatitis C. Subjects with undetectable HBV DNA or HCV RNA after anti-virus treatment can be enrolled;
3. HIV positive;
4. Other active infections of clinical significance;
5. Subjects with the following previous or accompanying diseases:

   • Subjects diagnosed as severe autoimmune diseases that require long term (more than 2 months) treatment with systemic immunosuppressants (steroids), or diseases with immune-mediated symptoms, including ulcerative colitis, Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus (SLE), and autoimmune vasculitis (e.g. Wegena granuloma);
6. Patients with previous diagnosis as motor neuron disease caused by autoimmunity;
7. Patients previously suffered from toxic epidermal necrolysis (TEN)
8. Patients with any mental illness, including dementia, mental changes, which may cause difficulties understanding the informed consent and related questionnaires;
9. Patients with serious uncontrollable diseases, which may interfere with the therapies in this study;
10. Patients with other active malignancies in the past 5 years excluding those with completely cured basal or squamous skin cancers, superficial bladder cancers or primary breast cancers without need of follow-up treatment;
11. Subjects receiving systemic steroids or steroid inhalants;
12. Patients who have received tumor immunotherapy (including monoclonal antibody against PD-1, PD-L1, PD-L2, CD137 or CTLA-4, or cell therapy) in the past 4 weeks;
13. Subjects allergic to immunotherapies or related drugs;
14. Patients with metastatic lesions in meninges or central nervous system, or clear evidence of central nervous system diseases with continuous significant symptoms in the last 6 months;
15. Patients with NYHA class II heart failure, or hypertension incontrollable by standard care, or medical history of myocarditis, or heart attack within a year;
16. Subjects who have received or are going to receive organ transplantation;
17. Patients with active bleeding;
18. Patients with incontrollable pleural or abdominal fluid that needs clinical treatment or intervention;
19. Patients as determined by the investigators to be inappropriate for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
DLT | 28 days following infusion
  To assess the safety and tolerability of CCT301-38 cell therapy for patients with AXL-positive (IHC 1+ or greater in ≥50% tumor cells) relapsed or refractory sarcomas.

SECONDARY OUTCOMES:
ORR | Up to 52 weeks
  Proportion of subjects with the best overall response (BOR) of subjects with PR (partial response) and CR (complete response) as determined by local investigator using RECIST 1.1
DCR | Up to 52 weeks
  Disease control rate: The proportion of subjects with CR (complete response), PR (partial response) or SD (stable disease lasting over 6 months) as determined by local investigator using RECIST 1.1.
DOR | Up to 52 weeks
  Duration of response: The duration of time from record of response to first progression of disease as determined by RECIST 1.1 or death date not relevant to disease progression.
PFS | Up to 52 weeks
  Progression free survival: The time of disease progression by RECIST 1.1 or death since cell infusion.
TEAE | Up to 52 weeks
  Number, severity and duration of treatment of emergent adverse events (TEAEs) that occur during treatment according to NCI-CTCAE v 5.0.
PK | Up to 52 weeks
  The % of patients with detectable CCT301-38 cells in peripheral blood. [Time Frame: Up to 52 weeks]
Biomarker | Up to 52 weeks
  To evaluate the correlation of AXL biopsy score to ORR. [Time Frame: Up to 52 weeks]

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China